CLINICAL TRIAL: NCT07246161
Title: Detection of Orally Delivered Probiotic Strains in the Vaginal Microbiome of Healthy Female Adults
Brief Title: Vaginal Detection of Orally Delivered Probiotic Strains in Healthy Women
Acronym: VSS2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: L-032; 25AQ-1030 (Other: CRO Study Number. Evalulab)
Record Dates: First submitted 2025-11-13; First posted 2025-11-24 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Focus is on Healthy Subjects
Keywords: Probiotics; Women's Health

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental)
  Interventions: Other: Probiotic Formula 1
- Group 2 (Experimental)
  Interventions: Other: Probiotic Formula 2
- Group 3 (Experimental)
  Interventions: Other: Probiotic Formula 3

INTERVENTIONS:
Other: Probiotic Formula 1 — Includes 2 different probiotic strains differing from other intervention groups.
  Arms: Group 1
Other: Probiotic Formula 2 — Includes 2 different probiotic strains differing from other intervention groups.
  Arms: Group 2
Other: Probiotic Formula 3 — Includes 2 different probiotic strains differing from other intervention groups.
  Arms: Group 3

SUMMARY:
The purpose of the present study is to obtain more information on the transit of orally ingested probiotics to the vagina.

DETAILED DESCRIPTION:
Probiotics have emerged as novel supplements to support women's health, demonstrating benefits in maintain vaginal health and promoting recovery from dysbiosis. This includes various oral and vaginal probiotics shown to alleviate symptoms and enhance the reversal of vaginal dysbiosis.

Oral delivered probiotic strains suggest their ability to migrate and colonize the vagina to support vaginal health but is not well understood. Therefore, this study will aim to provide additional information on their transit to the vagina.

ELIGIBILITY:
Inclusion Criteria:

* Clinically healthy female between the ages of 18 and 50 years, inclusive,
* have a regular or predictable menstrual cycle
* Typically have regular bowel movements,
* Willing and able to consume a probiotic supplement for 4 weeks,
* Willing to discontinue consumption of probiotic supplement and probiotic-fortified products 2 weeks before the start of the study and throughout the study,
* Willing to discontinue fiber supplements 2 weeks before the start of the study, and throughout the study,
* Willing to provide 1 stool sample 4 times throughout the study,
* Willing to provide 2 vaginal swabs 4 times throughout the study,
* Willing to undergo vaginal pH swab measurements (with a swab) 5 times throughout the study,
* Willing to provide 2 perineal skin swabs (skin between the vagina and the anus) 3 times throughout the study,
* Willing to complete a pregnancy test at the screening visit.

Exclusion Criteria:

* Menopausal women,
* Vaginal pH < 2 or > 5 measured at screening,

  •. Menstruation during the sample collection times,
* Women that are lactating, pregnant, attempting to get pregnant, or have a positive pregnancy test,
* Use of vaginal probiotics in the last 3 months,
* Use of local vaginal antibiotics or antifungals in the last 3 months.
* Use of oral antibiotics or antifungals in the last month,
* Ongoing symptoms of vaginal and/or urinary tract infections,
* Current treatment for vaginal sepsis or urosepsis,
* Currently being treated for a severe chronic disease (e.g. cancer, renal failure, chronic inflammatory digestive or gastro-intestinal disease, immunodeficiency, etc.),
* Clinical diagnosis of a gynecological disease or condition (e.g, fibroma, endometriosis, polycystic ovarian syndrome, etc.),
* Clinical diagnosis of secondary dysmenorrhea,
* Intolerance, allergy or sensitivity to milk, soy, or yeast.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of probiotic stains in vaginal swabs after 28 days of oral intake | 28 days of oral intake

SECONDARY OUTCOMES:
Presence or absence of the probiotic stains in the vaginal swabs at days 0 & 14 of oral intake, and 1 week after the end of intervention (Day 35) | From enrollment to day 35
Presence or absence of the probiotic strains in perineal skin swabs at days 0, 14, and 28 of oral intake. | From enrollment to the 28th day.
Presence or absence of the probiotic strains in stool samples at days 0, 14 and 28 of oral intake. | From enrollment to 28th day
Viability of the probiotic strains recovered from vaginal swabs at days 0, 14, and 28 of oral intake, and 1 week after the end of the intervention (Day 35) | From enrollment to the 35th day.
Viability of the probiotic strains recovered from perineal skin swabs at day 0, 14, and 28 of oral intake. | From enrollment to 28th day
Changes in vaginal pH from baseline to 1 week after the end of the intervention (Day 35) | From baseline to day 35.
Changes in the abundance of endogenous and pathogenic bacterial and fungal species in the vagina at days 0, 14, 28 and 35. | From enrollment to the 35th day

OTHER OUTCOMES:
Number of adverse events (AEs) and serious adverse events (SAEs) reported throughout the study. | From enrollment to the 35th day

CONTACTS AND LOCATIONS:
Locations (1):
- Evalulab, Montreal, Canada